CLINICAL TRIAL: NCT05755113
Title: A Phase IIa Open Label Study Evaluating the Preliminary Efficacy of Intratumoural Tigilanol Tiglate in Advanced and/or Metastatic Soft Tissue Sarcoma of the Extremities and Body Wall.
Brief Title: A Clinical Study to Investigate the Efficacy of Intratumoral Tigilanol Tiglate in Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: QBiotics Group Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QB46C-H07; U1111-1282-2967 (Other: [WHO Universal Trial Number (UTN)])
Record Dates: First submitted 2023-02-16; First posted 2023-03-06 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Soft Tissue Sarcoma
Keywords: extremeties; body wall; advanced; metastatic
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis | interventions — EBC-46

STUDY DESIGN:
Intervention Model Description: Open label, single arm. Stage 1 - 10 evaluable participants, max of 5 treatments, 28 days apart. Stage 2 - up to 40 evaluable participants with a maximum of 10 participants in each of four histologically different groups: (i) angiosarcoma, (ii) leiomyosarcoma, (iii) myxofibrosarcoma, and (iv) other mixed origin sarcomas, max of 3 treatments, 7 days apart.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm, Open Label (Experimental): Single or multiple Intratumoural injections of tigilanol tiglate at up to a fixed dose of 3.6 mg/m2 (Body Surface Area [BSA]) per treatment.
  Interventions: Drug: Tigilanol Tiglate

INTERVENTIONS:
Drug: Tigilanol Tiglate — Tigilanol tiglate is a novel, short-chain diterpene ester in clinical development for intratumoural treatment of a wide range of solid tumours.
  Other Names: EBC-46

SUMMARY:
A Phase IIa open label study evaluating the preliminary efficacy of intratumoural tigilanol tiglate in advanced and/or metastatic soft tissue sarcoma of the extremities and body wall.

DETAILED DESCRIPTION:
Primary Objective

1. To evaluate tumour ablation in tumours and/or tumour segments following one or more treatments with tigilanol tiglate; and
2. To evaluate the effect of tigilanol tiglate on overall disease control (not limited to injected tumours) (Stage 2 only).

Secondary Objective

1. To assess the safety and tolerability of intratumoural injections with tigilanol tiglate; and
2. To evaluate systemic exposure through pharmacokinetic (PK) assessment after a single intratumoural injection of tigilanol tiglate.

Exploratory Objectives

1. To evaluate the microenvironment of injected tumours +/- non-injected tumours;
2. To evaluate the degree of immune response elicited with intratumoural tigilanol tiglate;
3. To evaluate local recurrence rate; and
4. To evaluate metabolites after a single intratumoural injection of tigilanol tiglate (Stage 2 only).

ELIGIBILITY:
Inclusion Criteria:

1. Are willing and able to provide written informed consent for the study prior to any protocol-specific procedures and to comply with all local and study requirements.
2. Are ≥ 18 years of age on the day of providing informed consent.
3. Have advanced and/or metastatic disease of the body wall or extremities that is amenable to intratumoural injection either by palpation or under ultrasound guided injection, that has been histologically or pathologically confirmed as an STS. STS located on the scalp may also be considered for treatment.
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
5. Have life expectancy of more than 12 weeks.
6. Have adequate renal and hepatic function as assessed by the Investigator.
7. Female participants who are Women Of Child-Bearing Potential (WOCBP) must have a negative serum pregnancy test at Screening (within 14 days of the first study drug administration), must be willing to use a highly effective contraception from date of consent, throughout the study period and up to 30 days after the last study drug administration, and must not be breastfeeding.
8. Male participants with a potentially fertile female partner are eligible if they have had a vasectomy or are willing to use adequate contraception from prior to commencement of study drug administration, throughout the study period and up to 30 days after the last study drug administration, and must not donate sperm throughout the study period and up to 30 days after the last study drug administration.

Exclusion Criteria:

1. Are planning to receive intratumoural treatment or radiotherapy to any of the tumours intended for injection within 28 days prior to Screening, or during treatment with tigilanol tiglate.
2. Have a tumour intended for injection that is immediately adjacent to, or with infiltration into, any major artery or vein (e.g., if the tumour for injection is located adjacent to the jugular vein).
3. Are receiving or have received other investigational agents or have used an investigational device without undergoing a 28-day (or 5 half-lives, whichever is shorter) wash-out period prior to their first treatment with tigilanol tiglate. These patients must have recovered from all AEs due to previous investigational therapies to ≤ Grade 1 at baseline.
4. Are receiving or have received systemic anticancer therapy, without undergoing a 28-day (or 5 half-lives, whichever is shorter) wash-out period prior to their first treatment with tigilanol tiglate. These patients must have recovered from all AEs due to previous therapies to ≤ Grade 1 at baseline. Patients with ≤ Grade 2 neuropathy may be eligible following discussion with Sponsor Medical Monitor.
5. Have had major surgery within 28 days of their first treatment with tigilanol tiglate or anticipate the need for major surgery during the study period. Minor surgical procedures are permitted, but with sufficient time for wound healing.
6. Have known, active brain metastases and/or carcinomatous meningitis. Participants who have previously treated brain metastases and are neurologically stable can be included.
7. Have any bleeding diathesis or coagulopathy that would make intratumoural injection or biopsy unsafe, or if they are on therapeutic warfarin therapy.
8. Have a history of allergic reactions or severe hypersensitivity (Grade ≥ 3) attributed to tigilanol tiglate or compounds of similar chemical or biologic composition to tigilanol tiglate, any of its excipients or other agents used in the study.
9. In the opinion of the treating Investigator, they are not an appropriate candidate for the study for any reason (e.g., they have known psychiatric or substance abuse disorder that would interfere with their ability to cooperate with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Tumour Response | 6 months
  Proportion of participants who have achieved partial or complete ablation of treated tumour(s) and/or tumour segment(s) following injection(s) with tigilanol tiglate.
ORR as determined by RECIST | 3 and 6 months post initial treatment (Stage 2 only)
  Objective Response Rate (ORR) as Determined by Response Evaluation Criteria in Solid Tumours (RECIST) V1.1

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 6 months
  Total number of Adverse Events (AEs) and Serious Adverse Events (SAEs) and number of AEs and SAEs deemed related to tigilanol tiglate.
Systemic Exposure | Up to 24 hours after the first dose
  Evaluation of how much tigilanol tiglate is circulating in the blood after a single injection.

OTHER OUTCOMES:
Tumour Microenvironment | 7 days before and between 28 and 56 days after standard of care (Stage 2).
  To assess changes in the tumour microenvironment by looking at the change from baseline of immune cell infiltration in tumour biopsy tissue collected from injected and/or non-injected tumours after injection with tigilanol tiglate.
Evaluation of Peripheral Blood Mononucleocytes (PBMCs) | 24 weeks
  Evaluation of Peripheral Blood Mononucleocytes (PBMCs).
Local Recurrence Rate at injection site(s) | 6 months
  Percentage of participants with local recurrence at injection site(s) at 6-months after first treatment.
Metabolite analysis | 24hrs following first injection.
  Metabolite analysis following a single intratumoural injection of tigilanol tiglate (Stage 2 only).

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Bartlett, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Centre, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No